CLINICAL TRIAL: NCT05505630
Title: The Effects of Sedatives on Tobacco Use Disorder Version 2
Acronym: SED-TUD2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Nida Addiction Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00081012; 10595 (Other: Nida Addiction Research Center)
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Smoking
Keywords: nicotine addiction; smoking; placebo; sedatives
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use Disorder; Smoking | interventions — Ketamine; Neoadjuvant Therapy; Midazolam; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Saline first injection; ketamine second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of placebo at the first injection visit and a single intravenous infusion ketamine at the second injection visit.
  Interventions: Drug: Ketamine; Drug: Saline
- Saline first injection; midazolam second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of placebo at the first injection visit and a single intravenous infusion midazolam at the second injection visit
  Interventions: Drug: Midazolam; Drug: Saline
- Saline first injection; dexmedetomidine second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of placebo at the first injection visit and a single intravenous infusion dexmedetomidine at the second injection visit.
  Interventions: Drug: Dexmedetomidine; Drug: Saline
- Ketamine first injection; Saline second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of ketamine at the first injection visit and a single intravenous infusion placebo at the second injection visit.
  Interventions: Drug: Ketamine; Drug: Saline
- Ketamine first injection; midazolam second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of ketamine at the first injection visit and a single intravenous infusion midazolam at the second injection visit.
  Interventions: Drug: Ketamine; Drug: Midazolam
- Ketamine first injection; dexmedetomidine second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of ketamine at the first injection visit and a single intravenous infusion dexmedetomidine at the second injection visit.
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine
- Midazolam first injection; Saline second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of midazolam at the first injection visit and a single intravenous infusion placebo at the second injection visit.
  Interventions: Drug: Midazolam; Drug: Saline
- Midazolam first injection; ketamine second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of midazolam at the first injection visit and a single intravenous infusion ketamine at the second injection visit.
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam first injection; dexmedetomidine second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of midazolam at the first injection visit and a single intravenous infusion dexmedetomidine at the second injection visit.
  Interventions: Drug: Midazolam; Drug: Dexmedetomidine
- Dexmedetomidine first injection; Saline second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of dexmedetomidine at the first injection visit and a single intravenous infusion placebo at the second injection visit.
  Interventions: Drug: Dexmedetomidine; Drug: Saline
- Dexmedetomidine first injection; ketamine second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of dexmedetomidine at the first injection visit and a single intravenous infusion ketamine at the second injection visit.
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine
- Dexmedetomidine first injection; midazolam second injection (Experimental): Subjects in this arm will receive a single intravenous infusion of dexmedetomidine at the first injection visit and a single intravenous infusion midazolam at the second injection visit.
  Interventions: Drug: Midazolam; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketamine — A single dose of IV ketamine will be administered.
  Other Names: a dissociative anesthetic used medically for induction and maintenance of anesthesia
  Arms: Dexmedetomidine first injection; ketamine second injection; Ketamine first injection; Saline second injection; Ketamine first injection; dexmedetomidine second injection; Ketamine first injection; midazolam second injection; Midazolam first injection; ketamine second injection; Saline first injection; ketamine second injection
Drug: Midazolam — A single dose of IV midazolam will be administered
  Other Names: benzodiazepine medication
  Arms: Dexmedetomidine first injection; midazolam second injection; Ketamine first injection; midazolam second injection; Midazolam first injection; Saline second injection; Midazolam first injection; dexmedetomidine second injection; Midazolam first injection; ketamine second injection; Saline first injection; midazolam second injection
Drug: Dexmedetomidine — A single dose of IV dexmedetomidine will be administered
  Other Names: benzodiazepine medication
  Arms: Dexmedetomidine first injection; Saline second injection; Dexmedetomidine first injection; ketamine second injection; Dexmedetomidine first injection; midazolam second injection; Ketamine first injection; dexmedetomidine second injection; Midazolam first injection; dexmedetomidine second injection; Saline first injection; dexmedetomidine second injection
Drug: Saline — A single dose of IV saline will be administered
  Arms: Dexmedetomidine first injection; Saline second injection; Ketamine first injection; Saline second injection; Midazolam first injection; Saline second injection; Saline first injection; dexmedetomidine second injection; Saline first injection; ketamine second injection; Saline first injection; midazolam second injection

SUMMARY:
Double-blind, placebo-controlled, randomized mechanistic clinical trial to test an intravenous dose of either ketamine, midazolam, dexmedetomidine, or a placebo (saline) on cigarette smoking behavior, craving, and neural effects.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled, randomized mechanistic clinical trial will test non-treatment seeking smokers with an intravenous infusion of ketamine (0.71 mg/kg), midazolam (0.025 mg/kg), dexmedetomidine (0.025 mg/kg), or placebo, at least 2 weeks apart. Participants will complete 7-day ecological momentary assessment (EMA) of daily craving, withdrawal, and smoking behavior before and after each infusion. They will be asked to abstain from tobacco/nicotine for twenty-four hours post-infusion to induce withdrawal symptoms and return to the lab the following day to complete measures of craving, withdrawal, an MRI scan, and smoking latency. After this study visit, participants will be allowed to smoke as usual for the rest of the EMA diary period. Physical and subjective effects and adverse effects will be closely monitored throughout.

ELIGIBILITY:
Inclusion Criteria:

* Smokes cigarettes daily for at least 2 years
* Afternoon expired breath carbon monoxide at least 5 ppm or morning urinary cotinine at least 100 ng/ml
* Negative urine drug screen for psychoactive drugs and negative breath alcohol

Exclusion Criteria:

* Have an unstable medical condition or stable medical condition that would interact with study drug or participation, including chronic pulmonary disease, coronary artery disease, current brain tumor, current increased intracranial pressure or impaired consciousness
* History of serious head trauma or neurological disorder (e.g., seizure disorder)
* Have any of the following: hypertension (i.e., systolic >140 mm Hg and/or diastolic >90 mm Hg on three separate measures; systolic >170 or diastolic > 110 on any occasion), pre-existing severe gastrointestinal narrowing (pathologic or iatrogenic).
* Use of drugs that would interact with study drug or increase risk of adverse events
* Among women, pregnancy or lactation

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Difference in craving between drug and placebo | 24-hours post infusion
  difference in self-reported craving for cigarettes after infusions
Difference in tobacco withdrawal symptoms | 24-hours post infusion
  difference in self-reported withdrawal symptoms after infusions
Difference in cigarette demand | 24-hours post infusion
  difference in self-reported cigarette demand after infusions
Number of cigarettes smoked ad lib | 24-hours post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A Addicott, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT05505630/ICF_000.pdf